CLINICAL TRIAL: NCT00962377
Title: Early Invasive Monitoring Attenuation Through Gene Expression (EIMAGE) Trial
Brief Title: A Comparison of AlloMap Molecular Testing and Traditional Biopsy-based Surveillance for Heart Transplant Rejection Early Post-transplantation
Acronym: EIMAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: XDx (Industry)
Responsible Party: Debbie Pieretti, Sr. Director Clinical Operations, XDx, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CA-0007
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-12

CONDITIONS: Graft Rejection; Heart Diseases
Keywords: molecular expression testing; right ventricular endomyocardial biopsy
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AlloMap Molecular testing (Other): Gene expression profiling in the monitoring of asymptomatic heart transplant patients for acute cellular rejection.
  Interventions: Procedure: AlloMap Molecular Testing
- Endomyocardial biopsy (Active Comparator): Right ventricular endomyocardial biopsy in the monitoring of asymptomatic heart transplant patients for acute cellular rejection
  Interventions: Procedure: Endomyocardial biopsy

INTERVENTIONS:
Procedure: Endomyocardial biopsy — Right ventricular endomyocardial biopsy in monitoring of asymptomatic heart transplant patients for acute cellular rejection
  Other Names: EMB
  Arms: Endomyocardial biopsy
Procedure: AlloMap Molecular Testing — Gene expression profiling in the monitoring of asymptomatic heart transplant patients for acute cellular rejection.
  Other Names: GEP
  Arms: AlloMap Molecular testing

SUMMARY:
This study is designed to evaluate the safety and efficacy of a peripheral blood mononuclear cell gene expression profiling method (AlloMap) in monitoring asymptomatic heart transplant patients for acute rejection beginning 2-6 months(≥ 55-185 days) after transplantation.

DETAILED DESCRIPTION:
Cardiac allograft rejection is experienced by 20-50% of patients at least once during the first year after cardiac transplantation under the present immunosuppression regimens. The standard for rejection surveillance has been the endomyocardial biopsy (EMB). However, EMB is invasive, causes morbidity, and is subject to sampling error and inter-observer variability.

Gene expression profiling (GEP), with its high negative predictive value (NPV) for acute cellular rejection (ACR), appears to be well suited to identify low-risk patients who can be safely managed without routine invasive endomyocardial biopsy (EMB).

The Invasive Monitoring Attenuation through Gene Expression (IMAGE) multicenter study was conducted between the years 2005-2009 and studied patients who were >6 months-5 years post transplant. The IMAGE study demonstrated that the clinical outcome of heart transplant patients managed with AlloMap® was noninferior to patients managed with EMB. The EIMAGE study expands the time window under study to include patients who are 2 months (≥ 55 days) post-transplant. This earlier time frame of study is the primary difference between the EIMAGE study and the IMAGE study.

ELIGIBILITY:
Inclusion Criteria:

1. Heart transplant recipients who are 2-6 months (≥55 days -185 days) post-transplant at the time of the first study surveillance visit
2. Age ≥ 18 years
3. Left ventricular ejection fraction ≥ 50% by Echocardiography, Multiple Gated Acquisition (MUGA) scan, or ventriculography at study entry (baseline / enrollment study)

Exclusion Criteria:

1. Any clinical signs of declining graft function:

   * Symptoms of Congestive Heart Failure (CHF) at the first study surveillance visit
   * Signs of decompensated heart failure, including the development of a new S3 gallop at the enrollment visit
   * Elevated right heart pressures with diminished cardiac index < 2.2 L/min/m2 that is new compared to a previous measurement within 2 months
   * Decrease in LVEF as measured by echocardiography: ≥ 25% compared to prior measurement within 2 months
2. Rejection therapy for biopsy-proven ISHLT Grade 3A or higher during the preceding 2 months
3. Prior or current evidence of antibody-mediated rejection (AMR). AMR is defined according to the ISHLT 2004 Guidelines as positive histology and immunopathology (either immunofluorescence or immunoperoxidase) staining for AMR
4. Major changes in immunosuppression therapy within previous 30 days (e.g., discontinuation of calcineurin inhibitors, switch from mycophenolate mofetil to sirolimus or vice versa)
5. Unable to give written informed consent
6. Patient receiving hematopoietic growth factors (e.g., Neupogen, Epogen) currently or during the previous 30 days
7. Patients receiving ≥ 20 mg/day of prednisone equivalent corticosteroids at the time of first study surveillance visit
8. Patient enrolled in a trial requiring routine surveillance endomyocardial biopsies
9. Patient received transfusion within preceding 4 weeks
10. Patients with end-stage renal disease requiring some form of renal replacement therapy (hemodialysis or peritoneal dialysis)
11. Pregnancy at the time of first study surveillance visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival and intravascular ultrasound (IVUS) measures | 1.5 years
  Event-Free Survival (EFS) is a composite of: the development of hemodynamic compromise with rejection, allograft dysfunction (hemodynamic compromise without histologically confirmed rejection), death from any cause, or re-transplantation.
  IVUS co-primary endpoint: maximal intimal thickness of the coronary arteries from baseline (measured at 6 weeks ± 30 days) to month 12 of ≥0.5mm, as measured by IVUS.

SECONDARY OUTCOMES:
Time from enrollment to death from any cause, and cause of death. | 1.5 years
Number of biopsies performed. | 1.5 years
Time from study enrollment to biopsy-related complications, as well as the number and type of biopsy-related complications. | 1.5 years
QOL responses as collected from the SF-12 form | Enrollment and one year post-transplant
Biopsy-related patient preferences satisfaction using a non-validated survey | Enrollment and one year post transplant
Objective measurements of cardiac function | 1.5 years
Gene expression profiling scores and immunosuppressant doses | 1.5 years
Number of rejection episodes. | 1.5 years
Utilization of AlloMap or biopsy to manage corticosteroid weaning between month 6 and month 12 post-transplant. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Upen Patil, MD, Study Director — XDx, Inc.
Locations (1):
- Cedars-Sinai Medical Center, Beverly Hills, California, United States

REFERENCES:
- [Background] Deng MC, Eisen HJ, Mehra MR, Billingham M, Marboe CC, Berry G, Kobashigawa J, Johnson FL, Starling RC, Murali S, Pauly DF, Baron H, Wohlgemuth JG, Woodward RN, Klingler TM, Walther D, Lal PG, Rosenberg S, Hunt S; CARGO Investigators. Noninvasive discrimination of rejection in cardiac allograft recipients using gene expression profiling. Am J Transplant. 2006 Jan;6(1):150-60. doi: 10.1111/j.1600-6143.2005.01175.x. PMID 16433769
- [Background] Starling RC, Pham M, Valantine H, Miller L, Eisen H, Rodriguez ER, Taylor DO, Yamani MH, Kobashigawa J, McCurry K, Marboe C, Mehra MR, Zuckerman A, Deng MC; Working Group on Molecular Testing in Cardiac Transplantation. Molecular testing in the management of cardiac transplant recipients: initial clinical experience. J Heart Lung Transplant. 2006 Dec;25(12):1389-95. doi: 10.1016/j.healun.2006.10.002. No abstract available. PMID 17178330
- [Background] Evans RW, Williams GE, Baron HM, Deng MC, Eisen HJ, Hunt SA, Khan MM, Kobashigawa JA, Marton EN, Mehra MR, Mital SR. The economic implications of noninvasive molecular testing for cardiac allograft rejection. Am J Transplant. 2005 Jun;5(6):1553-8. doi: 10.1111/j.1600-6143.2005.00869.x. PMID 15888068
- [Background] Marboe CC, Billingham M, Eisen H, Deng MC, Baron H, Mehra M, Hunt S, Wohlgemuth J, Mahmood I, Prentice J, Berry G. Nodular endocardial infiltrates (Quilty lesions) cause significant variability in diagnosis of ISHLT Grade 2 and 3A rejection in cardiac allograft recipients. J Heart Lung Transplant. 2005 Jul;24(7 Suppl):S219-26. doi: 10.1016/j.healun.2005.04.001. PMID 15993777
- [Result] Pham MX, Teuteberg JJ, Kfoury AG, Starling RC, Deng MC, Cappola TP, Kao A, Anderson AS, Cotts WG, Ewald GA, Baran DA, Bogaev RC, Elashoff B, Baron H, Yee J, Valantine HA; IMAGE Study Group. Gene-expression profiling for rejection surveillance after cardiac transplantation. N Engl J Med. 2010 May 20;362(20):1890-900. doi: 10.1056/NEJMoa0912965. Epub 2010 Apr 22. PMID 20413602
- See also: Information on molecular expression testing — http://www.xdx.com/allomap/
- See also: Sponsor's website — http://xdx.com/